CLINICAL TRIAL: NCT03777839
Title: Evaluation of 18F-Fluorodeoxyglucose Positron Emission Tomography Imaging in Myocarditis
Brief Title: PET-FDG in Myocarditis
Acronym: PETMYO
Status: Completed | Type: Observational
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Matthieu Pelletier-Galarneau, MD MSc, Adjunct Professor of Clinic, Montreal Heart Institute
Other Study IDs: 2019-2395
Record Dates: First submitted 2018-12-13; First posted 2018-12-17 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2023-10

CONDITIONS: Myocarditis; Viral Myocarditis
MeSH Terms: conditions — Myocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: FDG PET/CT — FDG PET CT imaging with rest perfusion imaging

SUMMARY:
This study evaluates the diagnostic performance of 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (FDG) positron emission tomography/computed tomography (PET/CT) with rest perfusion imaging for the diagnosis of myocarditis. Patients with clinical suspicion of myocarditis will be recruited and undergo a rest myocardial perfusion scan and a FDG PET/CT scan following a myocardial suppression protocol.

DETAILED DESCRIPTION:
Myocarditis is characterized by myocardial inflammation, which can lead to fibrosis and heart failure.

FDG PET/CT, with appropriate suppression protocol including high-fat-low-carbohydrate diet, fasting, and IV heparin, can be use to detect myocardial inflammation. It is frequently used for the diagnosis of inflammation in cardiac sarcoidosis. After the initial inflammatory phase, inflammation resolves and fibrosis can seen. Resting perfusion imaging will allow identification of fibrosis. The combination of FDG PET/CT and rest perfusion imaging could allow detection of the various phases of myocarditis; inflammation and fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Clinical suspicion of myocarditis due to findings such as:

   1. Symptoms and signs of myocarditis such as dyspnea, orthopnea, palpitation, and chest pain, without other identifiable cause
   2. New onset of cardiovascular symptoms with recent history of viral disease or previous myocarditis
   3. Unexplained new onset of left ventricular dysfunction
   4. Unexplained elevated troponin
   5. Magnetic resonance imaging findings suggestive of myocarditis, such as late gadolinium enhancement and edema
   6. Biopsy findings compatible with myocarditis
3. Women of childbearing potential must have a negative urine or blood pregnancy test
4. Capable of giving informed consent and the consent must be obtained prior to any study related procedures
5. Subject's with body mass index inferior or equal to 45 kg/m2

Exclusion Criteria:

1. Female subject who is pregnant or breastfeeding and unwilling to stop for 24h
2. Claustrophobia or inability to lie still in a supine position for imaging purposes
3. Unwillingness or inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 50 subjects with high clinical suspicion of myocarditis will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity of FDG PET/CT imaging with rest perfusion imaging to detect myocarditis | 1 year
  Sensitivity of FDG-PET/CT with rest perfusion imaging

SECONDARY OUTCOMES:
Specificity and accuracy of FDG-PET/CT with rest perfusion imaging to detect myocarditis | 1 year
  Specificity and accuracy of FDG-PET/CT with rest perfusion imaging
Left ventricular ejection fraction | 1 year
  The association between subjects' outcome and quantitative assessment of left ventricular inflammation and scar will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Matthieu Pelletier-Galarneau, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided